CLINICAL TRIAL: NCT02741362
Title: A Phase I-II Open- Label Study to Assess the Safety, Tolerability, and Preliminary Efficacy of a Single Intravenous Dose of Autologous Adipose Stem Cell (Adult Human) to Subjects With Refractory Rheumatoid Arthritis, Relapsing Systemic Lupus Erythematosus or Sharp's Syndrome
Brief Title: Safety and Efficacy of Adipose Derived Stem Cells in Refractory Rheumatoid Arthritis, Systemic Lupus Erythematosus or Sharp's Syndrome
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Primary Investigator no longer with institution
Sponsor: Arkansas Heart Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICMS-2015-51
Record Dates: First submitted 2016-04-06; First posted 2016-04-18 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Systemic Lupus Erythematosus; Rheumatoid Arthritis; Sharp's Syndrome
Keywords: Type III hypersensitivity autoimmune disease
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis, Rheumatoid; Mixed Connective Tissue Disease | interventions — Tissue Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ADSC arm (Experimental): Single intravenous administration of Stromal Vacsular Fraction (SVF) cells soinating Adipose Derived Stem Cells (ADSC) 6 week baseline data prior to the injection of ADSC will be collected. 6 week, 3 months and 6 months follow up data will be compared against baseline.
  Interventions: Other: Intravenous injection of Stromal Vascular Fraction Cells (SVF) containing ADSCs; Other: Lipoaspiration

INTERVENTIONS:
Other: Intravenous injection of Stromal Vascular Fraction Cells (SVF) containing ADSCs
  Other Names: Tissue transplant
Other: Lipoaspiration

SUMMARY:
This is a Phase I-II open- label single-dose study in subjects with significant refractory Rheumatoid Arthritis (RA), relapsing Systemic Lupus Erythematosus (SLE) or Sharp's Syndrome (SS).

This study will enroll a minimum of 20 subjects for RA, 20 subjects for SLE and 20 patients for SS. 6 week data of serum Tumor Necrosis Factor- alpha (TNFa), Interleukin- 6 (IL-6), C- Reactive Protein (CRP), Erythrocyte Sedimentation Rate (ESR), Cluster of Differentiation (CD)4 +CD25 + Forkhead box P3(Foxp3) + regulatory T cells, Disease Activity Score for 28 joints (DAS-28) score and pain score will be collected in all patients who are enrolled in the study for the RA group (Baseline and 6 weeks after). For the SLE group, Transforming Growth Factor- beta (TGF-β), TNFa, IL-6, Interleukin- 17 (IL-17), CD3+CD8-IL17A+ T helper-17 (Th17) cells, CD4+CD25+Foxp3+ regulatory T cells and the Systemic Lupus Erythematosus Quality of Life Questionnaire (SLEQoL) score will be collected in all the subjects of this group. SS group will undergo the assessments of RA and SLE. Prior to the stem cell treatment, the patient will be assessed for 6 weeks by all the previously mentioned markers. Then, patients will receive the infusion of stromal vascular fraction cells containing the adult adipose derived stem cells 'aADSC' (single intravenous dose). The disease- modifying anti-rheumatic drugs (DMARDs) or the standard SLE treatment will not be interrupted with the exception of systemic steroids (excluding minimal maintenance dose of one steroid) during the duration of the study. Follow up visits will take place at 6 weeks, 3 Months and 6 Months after the cell infusion. Safety will be monitored on an ongoing basis, and an interim safety review will be conducted by the Investigator(s) and Sponsor after the first 10 patients have been enrolled and treated in each group.

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females ≥18 years
2. Cognitive competitiveness.
3. Diagnosis of refractory RA (patient's poor response of 3 months of DMARDs determined and documented by a rheumatologist) ,diagnosis of relapsing SLE (more than 2 episodes in a year during optimal medical SLE therapy) or diagnosis of Sharp syndrome (Alarcon-Segovia's criteria: patients with U1 Ribonucleic protein (RNP) ≥ 1:1600, and three of the following: Swollen hands, Synovitis, Myositis, Raynauld's phenomenon, Acrosclerosis)
4. Life expectancy greater than 8 months
5. Ability to understand and provide signed informed consent, or have a designated legal guardian or spouse legally able and willing to make such decisions on the subject's behalf
6. Reasonable expectation that patient will receive standard post-treatment care and attend all scheduled safety follow-up visits
7. No changes in active pulmonary medications for heart failure during the two weeks prior enrollment.
8. Written informed consent

Exclusion Criteria:

1. Currently on systemic steroids (if chronic steroid therapy cannot be stopped, the patient will qualify if he/she is on a minimum maintenance dose per SLE, RA or SS guidelines of only one systemic steroid and constituting a bioequivalent to normal endogenous levels of that hormone).
2. Dementia.
3. Presence of immune deficiency.
4. Currently on NSAIDs, TNFa inhibitors, Calcium channel blockers or P2Y12 inhibitors
5. Complicated type 2 diabetes mellitus (presence of diabetic foot, advanced kidney disease or retinopathy).
6. History of cancer within the past 5 years.
7. Presence of any other clinically-significant medical condition, psychiatric condition, or laboratory abnormality, that in the judgment of the Investigator or Sponsor for which participation in the study would pose a safety risk to the subject
8. Participation in another study with an investigational drug or device within 3 weeks prior to treatment
9. History within the past year of drug or alcohol abuse.
10. Females known to be pregnant, lactating or having a positive pregnancy test (will be tested during screening) or planning to become pregnant during the study.
11. Inability to comply with the conditions of the protocol.
12. Porphyria.
13. Allergy to sodium citrate or any "caine" type of local anesthetic.
14. Patient scheduled for hospice care.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Frequency of Adverse Events (AE) and Serious Adverse Events (SAE) during a 6 month follow up period. | 6 Months

SECONDARY OUTCOMES:
Quality of Life Questionnaires for SLE/ RA | 6 Months
  SLEQoL score
Quality of Life Questionnaires for RA | 6 Months
  DAS-28 score
Blood Flow Cytometry for CD4+CD25+Foxp3+ regulatory T cells | 6 Months
  CD4+CD25+Foxp3+ regulatory T cells,
Blood Flow Cytometry for CD3+CD8-IL17A+TH17 cells | 6 Months
  CD3+CD8-IL17A+TH17 cells
Serum C- reactive protein (CRP) | 6 Months
  C- reactive protein (CRP)
Erythrocyte Sedimentation Rate (ESR) | 6 Months
  Erythrocyte Sedimentation Rate (ESR)
Serum Tumor Necrosis Factor- alpha (TNFa) | 6 Months
  Tumor Necrosis Factor- alpha (TNFa)
Serum Transforming Growth Factor- beta (TGFb) | 6 Months
  Transforming Growth Factor- beta (TGFb)
Serum Interleukin- 6 (IL-6) | 6 Months
  Interleukin- 6 (IL-6)
Serum Interleukin- 17 (IL-17) | 6 Months
  Interleukin- 17 (IL-17)

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Rodriguez, MD PhD, Principal Investigator — Arkansas Heart Hospital
Locations (1):
- Arkansas Heart Hospital, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang D, Huang S, Yuan X, Liang J, Xu R, Yao G, Feng X, Sun L. The regulation of the Treg/Th17 balance by mesenchymal stem cells in human systemic lupus erythematosus. Cell Mol Immunol. 2017 May;14(5):423-431. doi: 10.1038/cmi.2015.89. Epub 2015 Oct 5. PMID 26435067
- [Background] Sharp GC, Irvin WS, Tan EM, Gould RG, Holman HR. Mixed connective tissue disease--an apparently distinct rheumatic disease syndrome associated with a specific antibody to an extractable nuclear antigen (ENA). Am J Med. 1972 Feb;52(2):148-59. doi: 10.1016/0002-9343(72)90064-2. No abstract available. PMID 4621694
- [Background] Deng W, Chen W, Zhang Z, Huang S, Kong W, Sun Y, Tang X, Yao G, Feng X, Chen W, Sun L. Mesenchymal stem cells promote CD206 expression and phagocytic activity of macrophages through IL-6 in systemic lupus erythematosus. Clin Immunol. 2015 Dec;161(2):209-16. doi: 10.1016/j.clim.2015.07.011. Epub 2015 Jul 22. PMID 26209923
- [Background] Garimella MG, Kour S, Piprode V, Mittal M, Kumar A, Rani L, Pote ST, Mishra GC, Chattopadhyay N, Wani MR. Adipose-Derived Mesenchymal Stem Cells Prevent Systemic Bone Loss in Collagen-Induced Arthritis. J Immunol. 2015 Dec 1;195(11):5136-48. doi: 10.4049/jimmunol.1500332. Epub 2015 Nov 4. PMID 26538398
- [Background] Kamata Y, Iwamoto M, Muroi K, Minota S. Repeated local implantation of autologous peripheral blood mononuclear cells for the treatment of ischaemic digits in patients with connective tissue diseases. Rheumatology (Oxford). 2011 May;50(5):906-10. doi: 10.1093/rheumatology/keq389. Epub 2010 Dec 15. PMID 21169196